CLINICAL TRIAL: NCT03049722
Title: Clinical Investigation Plan for the AVOPT Data Collection
Brief Title: Clinical Investigation Plan for the AVOPT Data Collection Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik Canada Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AVOPT
Record Dates: First submitted 2016-03-14; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Cardiac Pacemaker, Artificial

ARMS (1):
- AVOPT Patient (Experimental)
  Interventions: Device: Pacemaker

INTERVENTIONS:
Device: Pacemaker

SUMMARY:
The purpose of this study is to collect clinical data for the development and evaluation of a new device feature for automatic AV-delay (AVD) optimization.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with an Evia DR(T) or Entovis DR(T) pacemaker
* Possessing 1st or 3rd degree AV block
* Implanted with Biotronik bipolar RA and RV leads
* Implantation date should be at least 4 months prior to this study

Exclusion Criteria:

* Patient is a minor (18 years old or younger)
* Patient is pregnant or breast-feeding
* Patient does not have the legal capacity to provide consent
* Patient has Mobitz type I or Mobitz type II heart block
* Patient has persistent supraventricular tachycardia (including atrial fibrillation) or ectopic beats.
* Patient is participating in other clinical studies during the clinical study
* Patient is strictly pacemaker dependent (physician discretion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Correlation analysis between measured PWD and optimal AVD. | Up to 6 hours
  Data analysis will be performed on the collected data to relate P wave duration (PWD) measured from the far field IEGM to the optimal AVD determined from the hemodynamic assessment.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Rouge Valley Centenary, Scarborough Village, Ontario
  - CHUS - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec